CLINICAL TRIAL: NCT00321893
Title: Randomized Phase II Trial of Budesonide Turbuhaler® 800 Micrograms/Twice Daily Versus Placebo in High-Risk Population With Undetermined Lung Nodules Detected at Screening Low Dose CT Scan
Brief Title: Budesonide in Treating Patients With Lung Nodules at High Risk of Developing Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCI-2014-02166; MDA-05-5-01; MDA-S262/505; MDA-2005-0953 (Other: MD Anderson Cancer Center (MDACC)); EUDRACT-2005-004614-32; CDR0000470861; NCI-2012-02113 (Registry Identifier: NCI's Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2014-10

CONDITIONS: Lung Cancer
Keywords: Small cell lung cancer; Non-small cell lung cancer; Budesonide; Entocort EC; Pulmicort Respules; Rhinocort aqua; Aerosol budesonide treatment; Smoking
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Smoking | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Budesonide (Experimental): Inhaled Budesonide 800 ug twice daily for 1 year
  Interventions: Drug: Budesonide
- Arm II: Placebo (Placebo Comparator): Inhaled placebo twice daily for 1 year
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Budesonide — Inhaled Budesonide 800 micrograms (ug) twice daily for one year.
  Other Names: Entocort EC; Pulmincort Respules; Rhinocort aqua
  Arms: Arm I: Budesonide
Other: Placebo — Inhaled placebo twice daily for one year.
  Arms: Arm II: Placebo

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of budesonide may keep lung cancer from forming in patients with lung nodules.

PURPOSE: This randomized phase II trial is studying how well inhalation budesonide works in treating patients with lung nodules who are at high risk of lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the effect, in terms of size and number reduction of computed tomography (CT) scan-detected undetermined lung nodules, in asymptomatic subjects with lung nodules at high-risk for developing lung cancer treated with inhaled budesonide vs placebo.

Secondary

* Compare average modification of nodule size and nodule number due to inhaled budesonide versus placebo.
* Correlate the modulation of biological markers of lung cancer in serum and sputum after treatment with the modification of lung nodules sizes.
* Determine treatment toxicity, side effects, and safety of inhaled budesonide.
* Evaluate the role of CT scans in estimating the grade of respiratory impairment and emphysema.
* Determine the effect of inhaled budesonide on respiratory function before and after treatment.

OUTLINE: This is a randomized, double-blind, placebo controlled study.

Participants are stratified according to gender, smoking habit (current vs former smoker), and nodule characteristics (solid vs semisolid or non-solid). Participants are randomized into 1 of 2 treatment arms.

* Arm I: Subjects receive inhaled budesonide twice daily for 1 year in the absence of unacceptable toxicity.
* Arm II: Subjects receive inhaled placebo twice daily for 1 year in the absence of unacceptable toxicity.

Participants undergo blood and sputum collection periodically during study for biomarker and correlative studies.

After completion of study therapy, subjects are followed at 1 month and continue CT scan screening.

PROJECTED ACCRUAL: A total of 202 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Current smokers or former smokers that have stopped within the last 15 years
2. Smoking history > 20 pack/years
3. Age > 50 years
4. Persistent lung nodules detected at Low dose computed tomography (LDCT) scan from previous year with 1 of the following:- longest diameter between 4&5 mm. Nodules may be stable or grown from the previous year (< 5 mm does not require additional diagnostic follow-up); longest diameter between 5.1 & 8 mm. Nodules may be stable or grown from the previous year. If grown, doubling time should be >1 year; longest diameter > 8 mm with negative PET scan, negative CT enhancement. Nodule should have grown with a doubling time between 1& 5 years; -longest diameter >8mm, non solid or partially solid nodules, stable or grown with doubling time between 1&5 years
5. Eastern Cooperative Oncology Group (ECOG) performance status < 1 (Karnofsky >60%)
6. Participants must have normal organ and marrow function as defined below: Leukocytes >3,000/mL, absolute neutrophil count greater than 1,500/mL, platelets greater than 100,000/mL, total bilirubin lower than 1.5 * upper normal institutional limits, aspartate aminotransferase (AST or SGOT)/alanine aminotransferase (ALT or SGPT) lower than 1.5 * upper normal institutional limits, creatinine lower than 1.5 * upper normal institutional limits
7. Females must be postmenopausal (ie, at least 1 year passed after the last menstruation), surgically sterile, or using acceptable contraceptive measures as judged by the Investigator. (A fertile woman is defined as being of child-bearing potential, from first menstruation to 1 year after last menstruation.). Negative serum beta-HCG for women of childbearing potential will be required at baseline. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. More than 6 lung nodules (suspect of chronic granulomatous disease)
2. Lung nodules with clearly benign morphological features at CT scan (i.e, homogenous calcification, solid nodules with regular and round or polygonal margins and distance from the pleura <1cm)
3. Subjects currently suffering from malignant disease or having had malignant disease within the last 5 years except for cervical carcinoma in situ and non melanoma skin cancer
4. Regular/chronic use of oral or inhaled corticosteroids; regular use being defined as a total of 3 months cumulative use in the last 12 months
5. Use of any other investigational agents at time of enrollment in the study during the three months preceding study enrollment
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to corticosteroid
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Any other factor that at the investigator's discretion contraindicates the use of inhaled corticosteroids
8. Pregnant or lactating females, or females planning to become pregnant during the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately. If needed, a pregnancy test will be performed on serum during baseline lab test
9. HIV-positive or other patients with immunodeficiencies should be excluded because of the risk of infections

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Veronesi, MD, Study Chair — European Institute of Oncology; Scott M. Lippman, MD, FACP, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Fumagalli C, Bianchi F, Raviele PR, Vacirca D, Bertalot G, Rampinelli C, Lazzeroni M, Bonanni B, Veronesi G, Fusco N, Barberis M, Guerini-Rocco E. Circulating and tissue biomarkers in early-stage non-small cell lung cancer. Ecancermedicalscience. 2017 Jan 31;11:717. doi: 10.3332/ecancer.2017.717. eCollection 2017. PMID 28194229
- [Derived] Veronesi G, Szabo E, Decensi A, Guerrieri-Gonzaga A, Bellomi M, Radice D, Ferretti S, Pelosi G, Lazzeroni M, Serrano D, Lippman SM, Spaggiari L, Nardi-Pantoli A, Harari S, Varricchio C, Bonanni B. Randomized phase II trial of inhaled budesonide versus placebo in high-risk individuals with CT screen-detected lung nodules. Cancer Prev Res (Phila). 2011 Jan;4(1):34-42. doi: 10.1158/1940-6207.CAPR-10-0182. Epub 2010 Dec 16. PMID 21163939
- [Derived] Lazzeroni M, Guerrieri-Gonzaga A, Serrano D, Varricchio MC, Veronesi G, Radice D, Feroce I, Nardi-Pantoli A, Lippman SM, Szabo E, Bonanni B. Budesonide versus placebo in high-risk population with screen-detected lung nodules: rationale, design and methodology. Contemp Clin Trials. 2010 Nov;31(6):612-9. doi: 10.1016/j.cct.2010.08.006. Epub 2010 Aug 16. PMID 20719253
- See also: University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 2006 to July 2007. Participants were recruited in Milan, Italy at the European Institute of Oncology.
Pre-assignment Details: Of 225 participants registered, 23 participants were excluded from the trial before assignment to groups.
Groups:
- Arm I: Budesonide: Inhaled Budesonide 800 micrograms (ug) twice daily for 1 year
Period: Overall Study
Arm/Group | Arm I: Budesonide | Arm II: Placebo
Started | 101 | 101
Completed | 77 | 87
Not Completed | 24 | 14
Not completed — Non-Compliance/Refusal | 16 | 10
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 6 | 3

BASELINE CHARACTERISTICS:
Population: Three (3) participants in Arm I: Budesonide, and one (1) in Arm II: Placebo later refused follow up CT and were excluded from overall analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Budesonide | Arm II: Placebo | Total
Number analyzed (Participants) | 101 | 101 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 94 | 190
  >=65 years | 5 | 7 | 12
Age, Continuous [Median (Full Range); unit: years] | 59 [52 to 72] | 59 [51 to 75] | 59 [51 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 78 | 79 | 157
Region of Enrollment [Number; unit: participants]
  Italy | 101 | 101 | 202

OUTCOME MEASURES:

1. Primary Outcome: Number CT- Detected Lung Nodules by Participant
Description: Lung nodules (nodule characteristics) in a person-specific analysis by Response Evaluation Criteria In Solid Tumors (RECIST) criteria using Computed Tomography (CT) detection: Persistent lung nodules detected at CT scan from previous year with 1 of following: longest diameter between 4&5 mm. Nodules may be stable or grown from the previous year (< 5 mm does not require additional diagnostic follow-up); longest diameter between 5.1& 8mm. Nodules may be stable or grown from the previous year. If grown, doubling time should be >1 year; longest diameter > 8 mm with negative positron positron emission tomography (PET) scan, negative CT enhancement. Nodule should have grown with doubling time between 1& 5 years; -longest diameter >8mm, non solid or partially solid nodules, stable or grown with doubling time between 1&5 years. Participants followed from baseline to 3 Years, follow up CT assessment planned at 12 months.
Time Frame: Baseline assessment
Population: Per person analysis in overall randomized study (202 participants) using identification (baseline) CT.
Measure: Number; unit: lung nodules
Units Other Than Participants: Lesions
Arm/Group | Arm I: Budesonide | Arm II: Placebo
Number analyzed (Participants) | 101 | 101
Number analyzed (Lesions) | 137 | 142
lung nodules
  Nonsolid | 12 | 14
  Partially Solid | 26 | 19
  Solid | 99 | 109

2. Primary Outcome: Size of CT- Detected Lung Nodules by Participant
Description: Lung nodules (nodule characteristics) in a person-specific analysis by Response Evaluation Criteria In Solid Tumors (RECIST) criteria using Computed Tomography (CT) detection. Nodule type categorized as: Nonsolid, Partially Solid, or Solid. Persistent lung nodules detected at CT scan from previous year with 1 of following: longest diameter between 4&5 mm. Nodules may be stable or grown from the previous year (< 5 mm does not require additional diagnostic follow-up); longest diameter between 5.1& 8mm. Nodules may be stable or grown from the previous year. If grown, doubling time should be >1 year; longest diameter > 8 mm with negative positron positron emission tomography (PET) scan, negative CT enhancement. Nodule should have grown with doubling time between 1& 5 years; -longest diameter >8mm, non solid or partially solid nodules, stable or grown with doubling time between 1&5 years
Time Frame: Baseline assessment
Population: Per person analysis. Per person analysis in overall randomized study (202 participants) using identification (baseline) CT.
Measure: Number; unit: lung nodules
Units Other Than Participants: nodules
Arm/Group | Arm I: Budesonide | Arm II: Placebo
Number analyzed (Participants) | 101 | 101
Number analyzed (nodules) | 137 | 142
lung nodules
  4-5 mm | 94 | 100
  5-8 mm | 40 | 42
  >8 mm | 3 | 0

3. Primary Outcome: Number of Participant Overall Responses as Measured by RECIST Criteria at 12 Months
Description: For single nodules >5 mm, clinical meaningful shrinkage of 30% or > longest diameter (LD) considered treatment success after 1 year treatment; for <5 mm, complete disappearance considered treatment success. Multiple lesions success is complete response (CR) or partial response (PR) according to RECIST while failure when progression disease (PD) or stable disease (SD). CR: disappearance all target & non target lesions + no appearance new lesions; PR: CR for target lesions+incomplete/SD for non target lesions+no new lesions or PR (i.e., 30%<sum LD target lesions) for target lesions + no PD for non target lesions + no appearance of new lesions; PD: PD (at least 20% > sum LD of target lesions) for target lesions irrespective of response of non target lesions or PD for non target lesions irrespective of response for target lesions/or appearance new lesions irrespective of response of target/or non target lesions; SD: neither sufficient shrinkage for PR nor increase for PD.
Time Frame: 12 Months
Population: Per person analysis. Excluded from analysis were three participants in Arm I: Budesonide and one participant in Arm II: Placebo who refused the Computed Tomography (CT) scan.
Measure: Number; unit: participants
Arm/Group | Arm I: Budesonide | Arm II: Placebo
Number analyzed (Participants) | 98 | 100
participants
  CR/PR | 2 | 1
  SD | 88 | 89
  PD | 8 | 10

4. Primary Outcome: Participant Overall Response (by Tumor Type Subsolid or Solid Tumor) as Measured by RECIST Criteria at 12 Months
Description: Number of participants with response according to RECIST criteria. For single nodules > 5 mm, clinical meaningful shrinkage of 30% or > of longest diameter (LD) considered treatment success after 1 year of treatment. For single nodules with LD <5 mm, complete disappearance considered treatment success. In case of multiple lesions success of treatment is when complete response (CR) or partial response (PR) occurs according to RECIST criteria.
Time Frame: 12 Months
Population: Per person analysis. Excluded from analysis were three participants in Arm I: Budesonide and one participant in Arm II: Placebo who refused the follow up Computed Tomography (CT) scan.
Measure: Number; unit: participants
Arm/Group | Arm I: Budesonide | Arm II: Placebo
Number analyzed (Participants) | 98 | 100
participants
  Subsolid, CR/PR | 2 | 1
  Subsolid, SD | 28 | 26
  Subsolid, PD | 3 | 3
  Solid, CR/PR | 0 | 0
  Solid, SD | 60 | 63
  Solid, PD | 5 | 7

ADVERSE EVENTS:
Time Frame: Adverse event collection at each visit from 3 month evaluation to month after follow up CT scan at 12 months, and with each visit. Overall active study period April 2006 to August 2008, 2 years and 4 months
Arm/Group | Arm I: Budesonide | Arm II: Placebo
Serious Adverse Events (participants affected / at risk) | 5/98 | 0/101
Other Adverse Events (participants affected / at risk) | 98/98 | 5/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Budesonide (N=98) | Arm II: Placebo (N=101)
Bipolar Affective Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Left Ureter Non-Invasive Carcinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostate Cancer (Renal and urinary disorders) | 1 (1) | 0 (0)
Surgery forArtery Stenosis Lower Limb (Vascular disorders) | 1 (1) | 0 (0)
TIA (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Budesonide (N=98) | Arm II: Placebo (N=101)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Ankle Trauma (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Asthmatic Attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
BPH (Renal and urinary disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 8 (8) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Candida (Infections and infestations) | 6 (7) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cervical Arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon Adenoma Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Conjunctival Hyperhemia (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 1 (1)
Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dental Abscess (Infections and infestations) | 7 (7) | 0 (0)
Dental Implant (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dental Surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Diabetic Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0)
Fever (General disorders) | 3 (3) | 0 (0)
Flu (General disorders) | 7 (12) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Pyrosis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hair Loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hands Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Hemorroids (Gastrointestinal disorders) | 1 (1) | 0 (0)
High ALT (Investigations) | 4 (4) | 0 (0)
High AST (Investigations) | 1 (1) | 0 (0)
High Bilirubin (Investigations) | 2 (2) | 0 (0)
High BUN (Investigations) | 3 (3) | 0 (0)
High Chloride (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
High Cholesterol (Investigations) | 2 (2) | 0 (0)
High Creatinine (Investigations) | 1 (1) | 0 (0)
High Leukocites (Investigations) | 1 (1) | 0 (0)
High Plasma Homocysteine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
High Potassium (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 0 (0)
Hot Flashes (Endocrine disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Inappetence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory Lung Lesion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Insect Bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Intercostal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee Distorsion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee Trauma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lipothymia (Nervous system disorders) | 1 (1) | 0 (0)
Loss of Memory (Nervous system disorders) | 1 (1) | 0 (0)
Low Cortisol (Endocrine disorders) | 15 (15) | 0 (0)
Low Hematocrit (Investigations) | 1 (1) | 1 (1)
Low Hemoglobin (Investigations) | 1 (1) | 0 (0)
Low Platelets (Investigations) | 1 (1) | 0 (0)
Low Voice (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 1 (1)
Lung Flogistic Lesion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Migratory Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pap Test Positivity (Infections and infestations) | 1 (1) | 1 (1)
Papilloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodonitis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Perleche (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Pharyngodynia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Prostatitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Retrosternal Weight (General disorders) | 1 (1) | 1 (1)
Rhinitis (Immune system disorders) | 2 (2) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scialorrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sciatic Neuralgia (Nervous system disorders) | 2 (2) | 0 (0)
Shoulder Dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Stipsis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Superventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Surgery for a Periumbelical Lipoma (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery for Suspect Oral Leukoplakia (Surgical and medical procedures) | 1 (1) | 0 (0)
Suspect Oral Luekoplakia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swallowing Difficulties (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Taste Alteration (Gastrointestinal disorders) | 8 (8) | 0 (0)
Teeth Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Teeth Sensitivity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Testis Cyst (Renal and urinary disorders) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Urine Frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Uterine Polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Vessel Injury-Artery: Lower Extremity (Vascular disorders) | 2 (2) | 0 (0)
Visus Reduction (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Weight Loss (Investigations) | 2 (2) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less